CLINICAL TRIAL: NCT00605410
Title: Duration of Protective Effect From Inhaled Ipratropium Bromide on Methacholine Airway Hyperresponsiveness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Dr. Donald W. Cockcroft, Department of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: BIO 07-161
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2008-07

CONDITIONS: Asthma
Keywords: Methacholine bronchoprovocation; Antimuscarinic
MeSH Terms: conditions — Asthma | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: ipratropium bromide
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ipratropium bromide — 2 puffs (40 micrograms) 2 puffs (0micrograms)
  Other Names: Atrovent HFA Inhalation Aerosol
  Arms: 1
Drug: placebo — Matched placebo
  Arms: 2

SUMMARY:
Certain lung disease medications can influence diagnostic tests and research investigations. This study will investigate how long ipratropium bromide must be withheld before a methacholine challenge test can be conducted. This information will be useful for validating current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma; stable and controlled
* FEV1 greater than or equal to 65% predicted

Exclusion Criteria:

* Concomitant lung disease other than asthma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
methacholine PC20 | 6hours and 12 hours post inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, Principal Investigator — Department of Medicine University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Illamperuma C, Davis BE, Fenton ME, Cockcroft DW. Duration of bronchoprotection of inhaled ipratropium against inhaled methacholine. Ann Allergy Asthma Immunol. 2009 May;102(5):438-9. doi: 10.1016/S1081-1206(10)60519-4. No abstract available. PMID 19496252